CLINICAL TRIAL: NCT01678326
Title: Endoscopic Ultrasound Guided Rendezvous or Direct Interventions Versus Advanced ERCP Techniques for Biliary Access and Therapy
Brief Title: EUS-Guided Rendezvous or Direct Interventions Versus Advanced ERCP Techniques for Biliary Access and Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Northwestern University (Other); University of Virginia (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Christopher Hemerski, Director of Luminal Oncology, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012.061-2-JSha
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Disorders of Gallbladder; Disorders of Biliary Tract
Keywords: Diseases Classified Elsewhere

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-Rendezvous or direct intervention (Active Comparator): EUS rendezvous or direct intervention involves: (1) using endoscopic-ultrasound technology to access the bile duct with a small needle and manipulate a wire across the biliary orifice and into the duodenum to be then retrieved endoscopically for ERCP (rendezvous ERCP), or (2) using endoscopic-ultrasound technology to directly puncture and perform intended biliary therapy
  Interventions: Procedure: EUS-Rendezvous or direct intervention
- Advanced ERCP Biliary Access Techniques (Active Comparator): Advanced ERCP techniques involve the following: precut access sphincterotomy and needle-knife fistulotomy. These are accepted techniques for biliary access in cases of difficult cannulation.
  Interventions: Procedure: Advanced ERCP Biliary Access Techniques

INTERVENTIONS:
Procedure: EUS-Rendezvous or direct intervention
  Arms: EUS-Rendezvous or direct intervention
Procedure: Advanced ERCP Biliary Access Techniques
  Arms: Advanced ERCP Biliary Access Techniques

SUMMARY:
The purpose of this study is to prospectively compare the efficacy of endoscopic ultrasound-guided biliary interventions (EUS-rendezvous or direct EUS-guided therapy) to that of advanced ERCP cannulation techniques in the setting of difficult cannulation. We hypothesize that EUS-guided interventions will be more successful and may be associated with the same complications as using advanced ERCP techniques in cases of difficult bile duct access.

DETAILED DESCRIPTION:
Background:

Biliary tract obstruction from stones or strictures are usually treated using endoscopic retrograde cholangiopancreatography (ERCP) techniques. However, biliary access (cannulation) during ERCP can be difficult. Overall cannulation success is about 90-95% at expert, centers. Difficult cannulation is associated with increased complication rates, as prolonged and repeated attempts can cause injury to the ampulla. When standard biliary cannulation fails advanced cannulation techniques, such as precut access sphincterotomy, are often indicated. These advanced techniques, however, increase the complication rate of ERCP, and still fail in a certain percentage of cases.

Endoscopic ultrasound-guided biliary interventions are relatively newer techniques that have emerged as a useful option to achieve biliary access or therapy when standard and advanced ERCP techniques for biliary access have failed. Many centers, including ours, are currently using EUS-guided interventions to facilitate ERCP access and therapy, when needed. EUS-guided interventions have emerged as a safe and effective procedure for gaining access to the biliary tree. A recent retrospective study comparing the safety and efficacy of EUS rendezvous to precut sphincterotomy (advanced ERCP technique for access), found that EUS-rendezvous was significantly more successful with no significant difference in the rate of procedural complications.

Currently, there are no accepted standards for deciding which biliary access technique to use in cases of difficult biliary cannulation. We hypothesize that EUS-guided biliary interventions will be more successful and may be associated with the same (or less) complications than using advanced ERCP techniques in cases of difficult bile duct access.

Procedures:

Patients referred for ERCP for biliary interventions at participating centers will be approached for consent. Patients who agree to participate will undergo a standard ERCP. The attending endoscopist will use standard ERCP techniques (i.e. cannulation with a standard cannula or sphincterotome with or without a wire) to gain biliary access for a minimum of ten minutes. If biliary access fails, the patient will be randomized to either the EUS-guided intervention arm or the advanced cannulation techniques arm of the study. The randomization ratio will be 50-50.

Methods of Data Analysis:

Based on current available data as well as our own experience, we estimated the success for immediate biliary access for EUS-guided intervention to be 90%, and for advanced ERCP cannulation techniques to be 75%. To detect this difference with power of 0.8 and a p-value of <0.05, a sample size of approximately 230 patients will be needed. Assuming that only 10% of patients that are consented will be randomized (based on the rationale that 90% of patients will either be successfully cannulated within 10 or will be excluded for other reasons) we estimate that approximately 2,300 patients will be consented for this study.

As this is the first study of its kind and it is possible that we will achieve statistical significance at an enrollment number earlier than our anticipated number of 230 participants two interim analyses are planned for this study. The first interim analysis is scheduled to occur after the enrollment of 70 patients (35 in each arm) and the second after enrollment of 140 patients (70 in each arm). The block randomization should result in equal numbers of patients in each arm at these enrollment levels. Adjustment for significance level at each interim analysis was calculated using the Pocock Boundary method (9). For either of the interim analyses, the level of significance required for termination of the trial for efficacy is p = 0.0221. An independent statistician will review the results and make recommendations regarding study termination based on results of interim analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed consent
* Patients referred to participating centers for ERCP with the intent to cannulate the bile duct for therapy

Exclusion Criteria:

* Patients with a bleeding diathesis (INR >1.4, platelets <80, current use of anticoagulant medications)
* Patients whose bile ducts are cannulated using standard methods
* Patients with prior biliary sphincterotomy or endoscopic papilla dilation
* Patients with previous surgical biliary-intestinal operations
* Patients with pancreas divisum
* Patients with indwelling pancreatic or biliary stent placement
* Patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2012-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Biliary access for therapy achieved (wire access across papilla or site of obstruction or wire access to enable successful therapy) | 24 hours
  Was the endoscopist able to achieve wire access into the biliary system in order to complete the intended therapy? Was intended therapy successful?

SECONDARY OUTCOMES:
Comparison of adverse events in the two arms. | Up to 1 month post procedure.
  Was there a difference in adverse events in the two arms. Adverse events include acute pancreatitis, hematoma, bile leak, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hamerski, M.D., Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Carr-Locke DL. Overview of the role of ERCP in the management of diseases of the biliary tract and the pancreas. Gastrointest Endosc. 2002 Dec;56(6 Suppl):S157-60. doi: 10.1067/mge.2002.129023. No abstract available. PMID 12447259
- [Background] Shah JN, Marson F, Weilert F, Bhat YM, Nguyen-Tang T, Shaw RE, Binmoeller KF. Single-operator, single-session EUS-guided anterograde cholangiopancreatography in failed ERCP or inaccessible papilla. Gastrointest Endosc. 2012 Jan;75(1):56-64. doi: 10.1016/j.gie.2011.08.032. Epub 2011 Oct 21. PMID 22018554
- [Background] Johnson GK, Geenen JE, Johanson JF, Sherman S, Hogan WJ, Cass O. Evaluation of post-ERCP pancreatitis: potential causes noted during controlled study of differing contrast media. Midwest Pancreaticobiliary Study Group. Gastrointest Endosc. 1997 Sep;46(3):217-22. doi: 10.1016/s0016-5107(97)70089-0. PMID 9378207
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Angsuwatcharakon P, Rerknimitr R, Ridtitid W, Ponauthai Y, Kullavanijaya P. Success rate and cannulation time between precut sphincterotomy and double-guidewire technique in truly difficult biliary cannulation. J Gastroenterol Hepatol. 2012 Feb;27(2):356-61. doi: 10.1111/j.1440-1746.2011.06927.x. PMID 21916994
- [Background] Masci E, Toti G, Mariani A, Curioni S, Lomazzi A, Dinelli M, Minoli G, Crosta C, Comin U, Fertitta A, Prada A, Passoni GR, Testoni PA. Complications of diagnostic and therapeutic ERCP: a prospective multicenter study. Am J Gastroenterol. 2001 Feb;96(2):417-23. doi: 10.1111/j.1572-0241.2001.03594.x. PMID 11232684
- [Background] Wang P, Li ZS, Liu F, Ren X, Lu NH, Fan ZN, Huang Q, Zhang X, He LP, Sun WS, Zhao Q, Shi RH, Tian ZB, Li YQ, Li W, Zhi FC. Risk factors for ERCP-related complications: a prospective multicenter study. Am J Gastroenterol. 2009 Jan;104(1):31-40. doi: 10.1038/ajg.2008.5. PMID 19098846
- [Background] Dhir V, Bhandari S, Bapat M, Maydeo A. Comparison of EUS-guided rendezvous and precut papillotomy techniques for biliary access (with videos). Gastrointest Endosc. 2012 Feb;75(2):354-9. doi: 10.1016/j.gie.2011.07.075. PMID 22248603